CLINICAL TRIAL: NCT01432938
Title: The Effect of Dulaglutide (LY2189265) on the Pharmacokinetics and Pharmacodynamics of Single Dose Warfarin in Healthy Subjects
Brief Title: A Study of the Effect of Dulaglutide on the Action of Warfarin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11549; H9X-MC-GBCS (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warfarin first, then Dulaglutide + Warfarin (Experimental): A single, 10-milligram (mg) dose of warfarin administered orally on Day 1 (Treatment 1). There was a washout period of at least 24 days between treatment periods. Then a single, 1.5-mg dose of dulaglutide administered subcutaneously on Day 1, followed by a single, 10-mg dose of warfarin administered orally on Day 3 (Treatment 2).
  Interventions: Biological: dulaglutide; Drug: Warfarin
- Dulaglutide + Warfarin first, then Warfarin (Experimental): A single, 1.5-mg subcutaneous dose of dulaglutide on Day 1, followed by a single, 10-mg oral dose of warfarin on Day 3 (Treatment 2). There was a washout period of at least 24 days between treatment periods. Then a single, 10-mg oral dose of warfarin on Day 1 (Treatment 1).
  Interventions: Biological: dulaglutide; Drug: Warfarin

INTERVENTIONS:
Biological: dulaglutide — Administered subcutaneously
  Other Names: LY2189265
Drug: Warfarin — Administered orally

SUMMARY:
Warfarin is a commonly used drug to prevent the blood from clotting. The purpose of this study is to determine if dulaglutide (LY2189265) affects how warfarin works. The study involves two different treatments (Treatment 1: warfarin; Treatment 2: dulaglutide + warfarin) separated by a minimum washout period of 24 days. In Treatment 1, the participant will receive 10 milligrams (mg) of warfarin on Day 1. In Treatment 2, the participant will receive a 1.5-mg dose of dulaglutide (LY2189265) as an injection on Day 1 and then a 10 mg dose of warfarin on Day 3. Participants will be randomly assigned into different treatment sequences. Participants in Treatment Sequence A will receive Treatment 1 then Treatment 2. Participants in Treatment Sequence B will receive Treatment 2 then Treatment 1.

ELIGIBILITY:
Inclusion Criteria:

* male participants with female partners of child-bearing potential, or partners who are pregnant or breastfeeding, agree to use a reliable method of contraception from the time of the first dose until 3 months after the last dose of investigational product, as determined by the investigator. The method may be one of the following:

  * condom with spermicidal agent
  * male participant sterilization
  * true abstinence (which is in line with the participant's usual lifestyle choice; withdrawal or calendar methods are not considered acceptable)
* female participants not of child-bearing potential and are postmenopausal or have undergone a documented hysterectomy (total or partial). Such participants will not be required to use contraception but must test negative for pregnancy at the time of enrolment. Postmenopausal is defined as at least 1 year post cessation of menses (without an alternative medical cause) with follicle stimulating hormone (FSH) ≥40 milli-international units per milliliter (mIU/mL)
* have a body mass index (BMI) of 18.5 to 32.0 kilograms per meter squared (kg/m^2), inclusive, at screening
* have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* have venous access sufficient to allow for blood sampling
* are reliable and willing to make themselves available for the duration of the study and are willing to follow study restrictions
* have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site

Exclusion Criteria:

* are currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* have known allergies to glucagon-like-peptide 1 (GLP-1)-related compounds including dulaglutide or to warfarin, related compounds, or any components of either formulation
* are persons who have previously completed or withdrawn from this study or any other study investigating dulaglutide in the 3 months prior to screening or have received glucagon-like peptides or incretin mimetics in the 3 months prior to screening
* history or presence of significant bleeding disorders that is, hematemesis, melena, severe or recurrent epistaxis, hemoptysis, hematuria, or intracranial hemorrhage
* have a personal history, family history, or current evidence of a bleeding disorder, coagulopathy, or clinically significant history of bleeding complications after surgical procedures, tooth extractions, nose or gingival bleeding, spontaneous bleeding (including bleeding into joint spaces)
* have a personal or family history of polycystic kidney disease or protein C or S deficiency
* have a history of major head trauma (with loss of consciousness) within the past year or minor head trauma (without loss of consciousness) within the last 3 months prior to screening
* have a history of or plan to undergo major surgery in the last 3 months prior to screening
* show positive for a fecal occult blood test at screening
* have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* have an abnormal blood pressure (after at least 5 minutes sitting) that, in the opinion of the investigator, increases the risks associated with participating in the study
* have a history or presence of cardiovascular, respiratory, hepatic, renal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis) or gastrointestinal disorder, for example relevant esophageal reflux or gall bladder disease, or any gastrointestinal disease which impacts gastric emptying (GE) (such as, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by GLP-1 analogs. Participants with mild dyslipidemia, and participants who had cholecystolithiasis (removal of gall stones) and/or cholecystectomy (removal of gall bladder) in the past, with no further sequelae, may be included in the study at the discretion of the screening physician
* Show evidence of significant active neuropsychiatric disease
* have family history of medullary thyroid cancer (MTC) or a genetic condition that predisposes to MTC
* regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* show evidence of hepatitis C and/or positive hepatitis C antibody
* show evidence of hepatitis B and/or positive hepatitis B surface antigen
* are women with a positive pregnancy test or women who are lactating
* have used or intend to use over-the-counter medication other than acetaminophen within 7 days prior to the first dose of warfarin or dulaglutide or prescription medication (with the exception of vitamin/mineral supplements and/or hormone replacement therapy [HRT]) within 14 days prior to dosing. Aspirin and other nonsteroidal anti-inflammatory drugs should not be taken from 2 weeks prior to the first dosing occasion
* show intended use of any drug or dietary supplement that may affect warfarin or coagulation within 14 days prior to the first dose of warfarin or dulaglutide or during the conduct of the study
* use or intended use of a drug that inhibits or induces cytochrome P450 (CYP)1A2, CYP2C9, CYP2C19, or CYP3A4 within 14 days prior to the first dose of warfarin or dulaglutide or during the conduct of the study
* have donated blood of more than 500 milliliters (mL) within the month prior to screening
* have an average weekly alcohol intake that exceeds 21 units per week (males up to age 65) and 14 units per week (males over 65 and females), or are unwilling to stop alcohol consumption from 48 hours prior to admission (Day -1 of the first treatment period) until discharge (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* are smokers
* have an international normalized ratio/prothrombin time (INR/PT) or activated partial thromboplastin time (aPTT) above the normal reference range at screening
* are females who menstruate
* have consumed grapefruit, cranberries, or grapefruit- or cranberry-containing products within 7 days prior to the first dose of warfarin or dulaglutide
* in the opinion of the investigator or sponsor, are unsuitable for inclusion in the study
* have any medical conditions, medical history or are taking any medication which are contraindicated within the warfarin Product Information Leaflet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

REFERENCES:
- [Derived] de la Pena A, Cui X, Geiser J, Loghin C. No Dose Adjustment is Recommended for Digoxin, Warfarin, Atorvastatin or a Combination Oral Contraceptive When Coadministered with Dulaglutide. Clin Pharmacokinet. 2017 Nov;56(11):1415-1427. doi: 10.1007/s40262-017-0531-7. PMID 28357715

RESULTS

PARTICIPANT FLOW:
Groups:
- Warfarin First, Then Dulaglutide + Warfarin: First Intervention: A single, 10-milligram (mg) dose of warfarin administered orally on Day 1 (Treatment 1).
  There was a washout period of at least 24 days between treatment periods.
  Second Intervention: A single, 1.5-mg subcutaneous dose of dulaglutide on Day 1, followed by a single, 10-mg dose of warfarin administered orally on Day 3 (Treatment 2).
- Dulaglutide + Warfarin First, Then Warfarin: First Intervention: A single, 1.5-mg subcutaneous dose of dulaglutide on Day 1, followed by a single, 10-mg dose of warfarin administered orally on Day 3 (Treatment 2).
  There was a washout period of at least 24 days between intervention periods.
  Second Intervention: A single, 10-mg dose of warfarin administered orally on Day 1 (Treatment 1).
Period: First Intervention
Arm/Group | Warfarin First, Then Dulaglutide + Warfarin | Dulaglutide + Warfarin First, Then Warfarin
Started | 14 | 14
Received at Least 1 Dose of Study Drug | 14 | 14
Completed | 12 | 14
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Washout Period of at Least 24 Days
Arm/Group | Warfarin First, Then Dulaglutide + Warfarin | Dulaglutide + Warfarin First, Then Warfarin
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Warfarin First, Then Dulaglutide + Warfarin | Dulaglutide + Warfarin First, Then Warfarin
Started | 12 | 14
Completed | 11 | 14
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study drug (dulaglutide or warfarin).
Groups:
- Entire Study Population: Participants who received at least one dose of study drug (dulaglutide or warfarin).
Arm/Group | Entire Study Population
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve (AUC) of R-warfarin and S-warfarin
Description: Area under the concentration versus time curve (AUC) from zero to infinity was determined from plasma concentrations of the S- and R- enantiomers of warfarin.
Time Frame: Predose (warfarin) and up to 144 hours postdose on Day 1 for Treatment 1 (warfarin alone) and on Day 3 for Treatment 2 (warfarin in combination with dulaglutide)
Population: Participants who received at least one dose of warfarin with evaluable warfarin concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms times hours per milliliter
Groups:
- Warfarin Alone: A single, 10-milligram (mg) dose of warfarin administered orally on Day 1 of Treatment 1.
- Dulaglutide + Warfarin: A single, 1.5-mg dose of dulaglutide administered subcutaneously on Day 1 of Treatment 2, followed by a single, 10-mg dose of warfarin administered orally on Day 3 of Treatment 2.
Arm/Group | Warfarin Alone | Dulaglutide + Warfarin
Number analyzed (Participants) | 28 | 25
nanograms times hours per milliliter
  S-warfarin | 19200 (24) | 18900 (22)
  R-warfarin | 33000 (25) | 32900 (24)

2. Primary Outcome: Pharmacokinetics: Maximum Observed Drug Concentration (Cmax) of R-warfarin and S-warfarin
Time Frame: as for outcome 1
Population: Participants who received at least one dose of warfarin with evaluable warfarin concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Warfarin Alone | Dulaglutide + Warfarin
Number analyzed (Participants) | 28 | 25
nanograms per milliliter (ng/mL)
  S-warfarin | 530 (19) | 414 (23)
  R-warfarin | 530 (18) | 451 (19)

3. Primary Outcome: Pharmacokinetics: Time to Maximum Concentration (Tmax) of R-warfarin and S-warfarin
Time Frame: as for outcome 1
Population: Participants who received at least one dose of warfarin with evaluable warfarin concentration data.
Measure: Median (Full Range); unit: hours
Arm/Group | Warfarin Alone | Dulaglutide + Warfarin
Number analyzed (Participants) | 28 | 25
hours
  S-warfarin | 2.00 [1.00 to 4.00] | 4.00 [1.00 to 24.02]
  R-warfarin | 2.00 [1.00 to 4.00] | 8.00 [2.00 to 24.02]

4. Secondary Outcome: Pharmacodynamics: Area Under the International Normalized Ratio Curve (AUCINR) of Warfarin
Description: AUCINR was assessed from venous blood samples collected to determine the response variable INR at predose and at pre-determined intervals after the administration of warfarin.
Time Frame: as for outcome 1
Population: Participants who received at least one dose of warfarin with evaluable warfarin INR data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin Alone | Dulaglutide + Warfarin
Number analyzed (Participants) | 28 | 25
ratio | 157 (5) | 161 (5)

5. Secondary Outcome: Pharmacodynamics: Maximum Observed International Normalized Ratio (INRmax) of Warfarin
Description: Observed INRmax was assessed from venous blood samples collected to determine the response variable INR at predose and at pre-determined intervals after the administration of warfarin.
Time Frame: as for outcome 1
Population: Participants who received at least 1 dose of warfarin with evaluable warfarin INR data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin Alone | Dulaglutide + Warfarin
Number analyzed (Participants) | 28 | 25
ratio | 1.24 (13) | 1.27 (15)

ADVERSE EVENTS:
Groups:
- Warfarin Alone: A single, 10-milligram (mg) dose administered orally on Day 1 of Treatment 1.
  Timeframe: Treatment 1
- Dulaglutide Alone: A single, 1.5-mg dose administered subcutaneously on Day 1 of Treatment 2.
  Timeframe: Day 1 to Day 3 before dosing of warfarin in Treatment 2
- Dulaglutide + Warfarin: A single, 1.5-mg dose of dulaglutide administered subcutaneously on Day 1 of Treatment 2, followed by a single, 10-mg dose of warfarin administered orally on Day 3 of Treatment 2
  Timeframe: After dosing of warfarin on Day 3 of Treatment 2
Arm/Group | Warfarin Alone | Dulaglutide Alone | Dulaglutide + Warfarin
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 3/28 | 5/26 | 4/25
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Warfarin Alone (N=28) | Dulaglutide Alone (N=26) | Dulaglutide + Warfarin (N=25)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days